CLINICAL TRIAL: NCT03577691
Title: Efficacy of a Decision Aid for Hydroxyurea(HU) in Sickle Cell Disease(SCD)
Brief Title: Efficacy of a Decision Aid for Hydroxyurea in Sickle Cell Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lakshmanan Krishnamurti, Professor, Emory University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00101669
Record Dates: First submitted 2018-06-28; First posted 2018-07-05 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Sickle Cell Disease
Keywords: Blood Disorders; Hydroxyurea (HU); Decision Aid
MeSH Terms: conditions — Anemia, Sickle Cell; Hematologic Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, randomized,controlled, unblinded study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training for use of web based Decision Aid (Experimental): Subjects will be provided access to the decision aid website and will receive a log-in identification, user password and url at time of consent and will be guided during a 30 minutes training session to use the website. They will ben be asked to continue to peruse the website at home to learn more about hydroxyurea. Participants in each group will be further randomized to 1) pretest surveys and posttest surveys; and 2)only posttest surveys
  Interventions: Other: Training for use of web based Decision Aid; Other: Pretest surveys and posttest surveys; Other: Only posttest surveys
- No training for use of web based Decision Aid (Placebo Comparator): Subjects will receive a log-in identification, user password and url at time of scheduled appointment for web access. They will not receive training but will be instructed to maneuver through the website and access the information pertaining to hydroxyurea and access the videos for the purposes of learning. Participants will be asked to peruse the website for 30 minutes at time of consent then to continue to access the website at home to learn about hydroxyurea treatment. Participants in each group will be further randomized to 1) pretest surveys and posttest surveys; and 2)only posttest surveys
  Interventions: Other: No training for use of web based Decision Aid; Other: Pretest surveys and posttest surveys; Other: Only posttest surveys

INTERVENTIONS:
Other: Training for use of web based Decision Aid — Subjects will be guided during a 30 minutes training session to use the website
  Arms: Training for use of web based Decision Aid
Other: No training for use of web based Decision Aid — Subjects will not be guided during a 30 minutes training session to use the website
  Arms: No training for use of web based Decision Aid
Other: Pretest surveys and posttest surveys — Subjects will be randomized to one of two groups initially: Those who do not receive training for the decision aid and those who are trained to navigate the decision aid. subjects in each group will be randomized to complete pre test and posttest surveys or only posttest surveys that will take 15 mts of time
Other: Only posttest surveys — Subjects will be randomized to one of two groups initially: Those who do not receive training for the decision aid and those who are trained to navigate the decision aid. subjects in each group will be randomized to complete pretest and posttest surveys or only posttest surveys.

SUMMARY:
The trial is a prospective, randomized study to determine the efficacy of training for use of a web based Decision Aid for Hydroxyurea(HU) usage among subjects with Sickle Cell Disease(SCD). Subjects are randomized primarily either to using a web based decision aid with training versus without training. Subjects in each group will be further randomized to 1) subjects receiving pretest surveys; and 2) subjects that do not receive pretest surveys.

DETAILED DESCRIPTION:
Hydroxyurea (HU) has been demonstrated to be efficacious in reducing complications such as vasocclusive pain crises and acute chest syndrome in children and adults with Sickle Cell Disease (SCD) and in improving survival in adults. It is also the only disease-modifying therapy and the only drug approved by the FDA for use in patients with SCD. However significant barriers remain in prescription and utilization of HU. Some of the barriers are under prescription and when prescribed, underutilization by patients. The majority of the reasons for underutilization by patients being fear of cancer or other side effects, concern about lack of efficacy, and unwillingness to take the medicine or come to clinic or pharmacy.

Decision aids are designed to help patients improve their knowledge of the options, achieve a more accurate perception of risk and benefits of treatment, participate actively in decision making, and make choices more in keeping with their values and preferences. Decision aids have been shown to be effective in providing greater knowledge; lower decisional conflict among the subjects. The web based decision aid is also likely to serve as a tool for clarification of patient values to themselves and to their healthcare providers. The web based decision aid, sickleoptions.org is a rather extensive and detailed website with information regarding sickle cell disease(SCD) complications and standard of care monitoring and management as well as the treatment options of hydroxyurea, Endari, chronic blood transfusion, and bone marrow transplant. It is necessary to assure user ability to navigate all of the elements of the site. The study wants to determine the efficacy of training for a web based Decision Aid for Hydroxyurea(HU) usage among subjects with Sickle Cell Disease(SCD) that are randomized to using a web based decision aid with training versus without training.

In the first phase of the study cognitive interviews will be conducted with 10-20 parents of patients with SCD or patients with SCD age > 18 years for development of training to navigate website. Interviews will be conducted in 5-subject iterative cycles to identify ease of usability and issues regarding navigation and usability to develop a training guide for website.

After consent, subjects will be asked to complete demographic questionnaires. Subjects will be randomized to either receive training or to not receive training to use the website. All subjects will be asked to spend about 30mts navigating the website after consent. Those who are randomized to receive training will be trained to use it during this time. Those who do not receive training will be asked to navigate through the site on their own. They may be randomized to complete 4 question surveys during this time. Not everyone will need to complete these surveys. This will take about 15 minutes. They will then be contacted each week for the next 3 weeks with a reminder to use the website. At week 4 they will complete 5 surveys over the phone. They may be randomized to complete a telephone interview. This interview will take about 30 to 45 minutes and will be audio recorded for transcription and analysis. Subjects will then be contacted every 3 months for 1 year to see if they made a decision about whether or not to start hydroxyurea for themselves (>18 yr-old subjects) or their child. These phone calls will take less than 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with sickle cell disease ages 18 to 80 years, inclusive Or parents of children (ages 9 months to <18 years) whose child has not started Hydroxyurea
* Patients who have made a past decision to not obtain treatment with Hydroxyurea or who have not obtained treatment with Hydroxyurea in past 12 months. Or parents of children who have made a past decision to not obtain treatment with Hydroxyurea or who have not obtained treatment with Hydroxyurea in the past 12 months.
* Patients or parents of children who's doctor identifies the patient/child as someone who should be on Hydroxyurea
* All participants will be able to comprehend English
* Subjects will have access to the internet from iPad, smart phone, or personal computer
* For the cognitive interviews participants will not be eligible to consider hydroxyurea as a treatment option

Exclusion Criteria:

* Patient who has already made a decision to begin and has started Hydroxyurea. Or parent who has already made a decision for their child to begin and the child has started Hydroxyurea.
* Participated in prior Decision Aid study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge Survey score to estimate the impact of use of the Decision Aid with training versus without training in improving knowledge regarding HydroxyUrea for Sickle Cell Disease | Baseline and 4 week follow up
  Subjects knowledge will be tested by using a knowledge Survey that was given at baseline and at 4 weeks follow up phone call. It is a 27 True, False or Unsure questionnaire that tests subjects knowledge of understanding risk for severe lung disease (pulmonary hypertension). This test is administered to both groups that are in turn randomized to to receive the pretest AND posttest or just the posttest surveys.

SECONDARY OUTCOMES:
Change in decisional conflict scale to estimate the impact of use of the Decision Aid with training versus without training aid on decisional conflict | Baseline and 4 week follow up
  The decisional conflict scale (DCS) measures personal perceptions of: uncertainty in choosing options; modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice. There are 16 questions with score value from 0=strongly agree to 4=strongly disagree. Scores range from 0(no decisional conflict) to 100 (extremely high decisional conflict)
Change in decision self efficacy scale to estimate the impact of use of the Decision Aid with training versus without training aid on decisional conflict | Baseline and 4 week follow up
  The decision self efficacy scale measures self confidence or belief in one's abilities in decision making, including shared decision making. There are 11 questions with score value from 0=not confident at all to 4=very confident. Scores range from 0(extremely low self efficacy) to 100 (extremely high self efficacy)
Change in Preparation for Decision Making Scale to estimate the impact of use of the Decision Aid with training versus without training aid on decisional conflict | Baseline and 4 week follow up
  The 'Preparation for Decision Making' scale assesses a patient's perception of how useful a decision aid or other decision support intervention is in preparing the respondent to communicate with their practitioner at a consultation focused on making a health decision.There are 10 questions with score value from 0=not at all to 5=a great deal. High scores indicate higher perceived level of preparation for decision making

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanan Krishnamurti, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Health System, Atlanta, Georgia
  - Hughes Spalding Children's Hospital, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia